CLINICAL TRIAL: NCT03899818
Title: Impiego Del Pallone Medicato Per il Trattamento di Piccoli Vasi Coronarici in Confronto Con Stent Medicato - Drug Eluting Balloon Efficacy for Small Coronary Vessel Disease Treatment
Brief Title: Drug Eluting Balloon Efficacy for Small Coronary Vessel Disease Treatment
Acronym: PICCOLETO II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatebenefratelli and Ophthalmic Hospital (Other)
Responsible Party: Principal Investigator, Bernardo Cortese, Principal Investigator, A.O. Fatebenefratelli Milano, Italy, Fatebenefratelli and Ophthalmic Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICCOLETO2
Record Dates: First submitted 2019-02-19; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
Keywords: small vessels; drug coated balloon
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new generation DEB (Other): drug-eluting balloon (DEB)
  Interventions: Device: drug-eluting balloon
- second generation DES (Other): standard therapy with second generation drug-eluting stent (DES)
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-eluting balloon — Patients will be randomized to drug-eluting balloon (DEB) or standard therapy with second generation drug-eluting stent (DES)
  Arms: new generation DEB
Device: drug-eluting stent — Patients will be randomized to drug-eluting balloon (DEB) or standard therapy with second generation drug-eluting stent (DES).
  Arms: second generation DES

SUMMARY:
This is a prospective, multicentre, randomized clinical study of consecutive patients with coronary artery disease in vessels with diameter ≤2.75 mm. Patients will be randomized to drug-eluting balloon (DEB) or standard therapy with second generation drug-eluting stent (DES). Study population will consist of 240 patients with stable or unstable angina

ELIGIBILITY:
Inclusion Criteria

1. Age >18 years.
2. Stable or unstable coronary artery disease.
3. Native coronary artery lesion in vessel with diameter <2.75 mm.
4. Clinical indication to percutaneous coronary intervention (PCI).

Exclusion criteria

1. Enrolment in another study with any investigational drug or device.
2. Acute or recent (≤48 hours) myocardial infarction.
3. Creatinine clearance <50 ml/min.
4. Left ventricle ejection fraction <30%.
5. Any known allergy, hypersensitivity or intolerance to any drug used during or after the procedure.
6. Heavily calcified and severely tortuous lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Verify the non-inferiority of DCB | up to 6 months
  the primary objective of the study is the non-inferiority of the DCB compared to DES in terms of absence of restenosis, defined as reoccurrence of stenoses of at least 50% of the lumen of the vessel at angiographic follow-up (6 months after surgery).

SECONDARY OUTCOMES:
Number of Participants with changes of vessels lumen | up to 12 months
  any differences between groups in terms of vascular changes to angiography.
Concentration in blood chemistry | up to 6 months
  changes of concentration in blood chemistry between the groups
Number of Participants with adverse events | up to 12 months
  appearance of major cardiovascular adverse events

REFERENCES:
- [Derived] Fezzi S, Trevisanello A, Buccheri D, Borgi M, Orrego PS, Zoccai GB, Cortese B. Physiological Performance of Drug-Coated Balloons in Small Coronary Arteries PICCOLETO II muFR. Catheter Cardiovasc Interv. 2025 Feb;105(3):643-649. doi: 10.1002/ccd.31376. Epub 2024 Dec 24. PMID 39718036
- [Derived] Cortese B, Testa G, Rivero F, Erriquez A, Alfonso F. Long-Term Outcome of Drug-Coated Balloon vs Drug-Eluting Stent for Small Coronary Vessels: PICCOLETO-II 3-Year Follow-Up. JACC Cardiovasc Interv. 2023 May 8;16(9):1054-1061. doi: 10.1016/j.jcin.2023.02.011. Epub 2023 Apr 19. PMID 37164603
- [Derived] Cortese B, Di Palma G, Guimaraes MG, Piraino D, Orrego PS, Buccheri D, Rivero F, Perotto A, Zambelli G, Alfonso F. Drug-Coated Balloon Versus Drug-Eluting Stent for Small Coronary Vessel Disease: PICCOLETO II Randomized Clinical Trial. JACC Cardiovasc Interv. 2020 Dec 28;13(24):2840-2849. doi: 10.1016/j.jcin.2020.08.035. Epub 2020 Nov 25. PMID 33248978